CLINICAL TRIAL: NCT05501275
Title: Evaluation of Life Quality in Post Stroke Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Palacky University (Other)
Responsible Party: Principal Investigator, Eva Prusova, Principal Investigator, Palacky University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: PalackyU
Record Dates: First submitted 2022-07-21; First posted 2022-08-15 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Stroke; Quality of Life
Keywords: stroke; life quality; evaluation
MeSH Terms: conditions — Stroke | interventions — Psychotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- With Psychoeducation (Experimental): interventional group will receive psychoeducation.
  Interventions: Behavioral: psychotherapy
- Basic Therapy Only (No Intervention): this group will receive only basic therapy

INTERVENTIONS:
Behavioral: psychotherapy — Psychotherapy and psychoeducation in patients after stroke.
  Arms: With Psychoeducation

SUMMARY:
Despite numerous advances in diagnosing procedures, treatment and prevention, stroke is considered a significant cause of long-term disability in the adult population Quality of life, which is deteriorated in patients after stroke (CVA), especially in the first years after stroke, is not only affected by the disease but is closely related to dignity and the satisfaction of human needs, including educational needs.

The term "Health-Related Quality of Life" (HRQoL) is used in the scientific literature as a criterion of change for medical purposes. It is an indicator of health service needs and a way to evaluate health status in a very efficient way. Psychoeducation can be applied in medical and nursing practice, as an intervention that can improve and/or maintain the quality of life, especially if it is provided to patients without a significant cognitive deficit. Psychoeducational programmes can be defined as didactic-therapeutic interventions that serve to provide information about the disease, emotional and social support and, last but not least, facilitate adaptation to new life situations.

DETAILED DESCRIPTION:
Detailed description:

The influence of selected aspects on HRQoL will be statistically assessed in the initial phase of the research. At a later stage, the monitored file will be randomized, in a predefined 1:1 ratio.

The control group will be provided only with conventional treatment focused on neurorehabilitation care according to the workplace's habits, and structured psychoeducation will be added to this usual care. The group psychoeducational interview, which reflects the issue of CVA, will be conducted face-to-face by a clinical psychologist, a health and social worker and a nurse. It will be limited by a 6-week therapy session 1 time per week, lasting approximately 45 minutes.

Patients will be tested with 6 standardized questionnaires in the Czech language version initially before the start of treatment and subsequently one month post the completion date of their treatment. The EuroQol-5 (EQ-5D-5L) instrument will be used to assess HRQoL. The Patient Dignity Inventory (PDI) questionnaire has been chosen to identify problems related to problems associated with patient dignity. The Mini-Mental State Examination (MMSE) cognitive test will be used to indicatively detect dementia and the Beck Depression Inventory Second Edition (BDI-II) will be used to diagnose the severity of depressive symptoms. The Visual Analogue Scale (VAS) will be used to objectify the perception of pain and the Barthel Index (BI) for scoring ADL. At the same time, selected relevant clinical and anamnestic data will be extracted from the medical records.

ELIGIBILITY:
Inclusion Criteria:

* adult with a clinical diagnosis of CVA in his/her medical history, lasting at ≥ 6 months and ≤ 3 years since the primo-attack,
* first hospitalized in a specialized medical institution,
* partial self-sufficiency,
* signed informed consent.

Exclusion Criteria:

* non-cooperation,
* recurrent CVA,
* severe depression with BDI-II score ≥ 40,
* dementia with MMSE score ≤ 25,
* presence of cancer and/or the end-stage of the disease.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 447 (Actual)
Dates: Start 2021-09-14 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Change in the Health-Related Quality of Life (HRQoL) in patients after stroke | 3 months
  Change in the Health-Related Quality of Life (HRQoL) [Time Frame: Baseline state (immediately prior to the rehabilitation facility admission) and follow-up monitoring (two and a half months after the rehabilitation facility admission)].
  Health-Related Quality of Life (HRQoL) is assessed using the European Quality of Life Questionnaire version 5, level 5 instrument. The output is an index (HRQoL dimension). Subsequently, the respondents are asked to indicate their subjectively perceived health condition.

SECONDARY OUTCOMES:
Change in patient´s dignity, level of depression, functional independence and pain | before the intervence and after 3 months
  Several scales were used:
  * to measure the patient´s dignity: Patient Dignity Inventory
  * to measure the level of depression: Beck Depression Inventory-II (BDI-II)
  * to measure the level of functional independence: Barthel Index (BI)
  * to measure the level of pain: visual analogue scale (VAS)

CONTACTS AND LOCATIONS:
Overall Officials: David Skoloudik, Prof, Principal Investigator — Faculty of Medicine, University of Ostrava, Syllabova 19, 703 00 Ostrava 3, Czech Republic
Locations (1):
- Palacky University, Olomouc, Czechia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hamid GM, MacKenzie MA. CE: Early Intervention in Patients with Poststroke Depression. Am J Nurs. 2017 Jul;117(7):32-40. doi: 10.1097/01.NAJ.0000520919.26724.9b. PMID 28594643
- [Result] Mavaddat N, Sadler E, Lim L, Williams K, Warburton E, Kinmonth AL, Mant J, Burt J, McKevitt C. Perceptions of self-rated health among stroke survivors: a qualitative study in the United Kingdom. BMC Geriatr. 2018 Apr 2;18(1):81. doi: 10.1186/s12877-018-0765-8. PMID 29609550
- [Result] Verberne DPJ, Kroese MEAL, Staals J, Ponds RWHM, van Heugten CM. Nurse-led stroke aftercare addressing long-term psychosocial outcome: a comparison to care-as-usual. Disabil Rehabil. 2022 Jun;44(12):2849-2857. doi: 10.1080/09638288.2020.1849417. Epub 2020 Nov 26. PMID 33242261
- [Result] Ostwald SK, Godwin KM, Cron SG, Kelley CP, Hersch G, Davis S. Home-based psychoeducational and mailed information programs for stroke-caregiving dyads post-discharge: a randomized trial. Disabil Rehabil. 2014;36(1):55-62. doi: 10.3109/09638288.2013.777806. Epub 2013 Apr 17. PMID 23594060
- [Result] Olukolade O, Osinowo HO. Efficacy of Cognitive Rehabilitation Therapy on Poststroke Depression among Survivors of First Stroke Attack in Ibadan, Nigeria. Behav Neurol. 2017;2017:4058124. doi: 10.1155/2017/4058124. Epub 2017 Jun 27. PMID 28720980
- [Result] Brouns B, van Bodegom-Vos L, de Kloet AJ, Tamminga SJ, Volker G, Berger MAM, Fiocco M, Goossens PH, Vliet Vlieland TPM, Meesters JJL. Effect of a comprehensive eRehabilitation intervention alongside conventional stroke rehabilitation on disability and health-related quality of life: A pre-post comparison. J Rehabil Med. 2021 Mar 5;53(3):jrm00161. doi: 10.2340/16501977-2785. PMID 33369683